CLINICAL TRIAL: NCT04706078
Title: Clinical and Radiographic Evaluation of a Cross-shaped Incision Technique to Thick-gingiva and Thin-gingiva Patients Treated With Implant-supported Fixed Prosthesis
Brief Title: Clinical and Radiographic Evaluation of a Cross-shaped Incision Technique
Status: Completed | Type: Observational
Sponsor: Wen Luo (Other)
Responsible Party: Sponsor-Investigator, Wen Luo, Associate Professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2009033
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Clinical and Radiographic Effect; Thick-gingiva; Implant; Thin Gingiva

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thick-gingiva group: After insertion of the probe into the facial aspect of the sulcus, the peri-implant biotype can be categorized as thick-gingiva (outline if the probe cannot be seen through the gingival)
- thin-gingiva group: After insertion of the probe into the facial aspect of the sulcus, the peri-implant biotype can be categorized as thin-gingiva (outline of the probe can be seen through the gingival)
  Interventions: Diagnostic Test: The biotype of gingival

INTERVENTIONS:
Diagnostic Test: The biotype of gingival — The biotype of gingival was also determined by periodontal probe.
  Groups: thin-gingiva group

SUMMARY:
To evaluate a cross-shaped incision technique to thick-gingiva and thin-gingiva patients treated with implant-supported fixed prosthesis.

DETAILED DESCRIPTION:
Objective: To evaluate a cross-shaped incision technique to thick-gingiva and thin-gingiva patients treated with implant-supported fixed prosthesis. Methods and Materials: 55 patients received cross-shaped incision were assigned into thick-gingiva group (29 cases) and thin-gingiva group (26 cases). Follow-up examination was carried out 3 and 12 months after final restoration. Clinical and radiographic evaluation including gingival papilla height, modified plaque index, modified sulcus bleeding index, periodontal depth, and crestal marginal bone level were utilized.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health, no chronic systemic diseases.
2. All subjects included in this study needed to have one missing premolar or molar teeth with adjacent natural teeth.
3. All subjects included in the study had been treated with one bone-level implant insertion in the premolar or molar region.

Exclusion Criteria:

1. Active periodontal infections.
2. Heavy smoking habit (>10 cigarettes per day).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study samples were comprised of patients who had been treated with one bone-level implant (Osstem, Korea) insertion in the first molar region. Fifty-five subjects were selected from the patients who came to the Department of Oral Implantology, West China Hospital of Stomatology, Sichuan University in China between June 2018 and June 2020.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
papilla height | Between June 2018 and June 2020.
  Presence/absence of papilla height was assessed visually
Modified Plaque Index (mPI) | Between June 2018 and June 2020.
  plaque accumulation around the marginal peri-implant tissue was assessed
Modified Sulcus Bleeding Index | Between June 2018 and June 2020.
  the bleeding tendency of the marginal peri-implant tissue was evaluated
Probing Depth (PD, in millimeters) | Between June 2018 and June 2020.
  PD was assessed at the mid-buccal, mid-oral, mesial and distal aspects of each implant with a standard periodontal probe, and final value was determined by the average of four aspects
Gingival margin level | Between June 2018 and June 2020.
  Gingival margin level was assessed by calculating the vertical distance between the most apical point of gingival margin at the buccal aspect of the crown and line connecting the peak of the adjacent mesial and distal natural teeth

SECONDARY OUTCOMES:
first bone-implant contact (fBIC) and implant shoulder (IS) | Between June 2018 and June 2020.
  the landmarks of first bone-implant contact (fBIC) and implant shoulder (IS) were used for measurements. fBIC-IS was defined as the vertical distance the first bone-implant contact to implant shoulder, and the distance was assessed at the mesial and distal aspect of implant, respectively. When the marginal crestal bone was located coronal to the IS, a positive (+) value was given, where a negative (-) value when located apically to the IS, the value was deemed as zero when IS and fBIC coincided.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [1] Du H, Gao M, Qi C, Liu S, Lin Y. Drug-induced gingival hyperplasia and scaffolds: they may be valuable for horizontal food impaction. Med Hypotheses 2010;74:984-5. [2] Bidra AS. Nonsurgical management of inflammatory periimplant disease caused by food impaction: a clinical report. J Prosthet Dent 2014;111:96-100. [3] Koori H, Morimoto K, Tsukiyama Y, Koyano K. Statistical analysis of the diachronic loss of interproximal contact between fixed implant prostheses and adjacent teeth. Int J Prosthodont 2010;23:535-40. [4] Gastaldo JF, Cury PR, Sendyk WR. Effect of the vertical and horizontal distances between adjacent implants and between a tooth and an implant on the incidence of interproximal papilla. J Periodontol 2004;75:1242-6. [5] Chow YC, Wang HL. Factors and techniques influencing peri-implant papillae. Implant Dent 2010;19:208-19. [6] Müller HP, Heinecke A, Schaller N, Eger T. Masticatory mucosa in subjects with different periodontal phenotypes. J Clin Periodontol 2000;27:621-6. [7] Yao JW, Wang HL. Assessment of Peri-implant Soft Tissue Adaptive Pressure and Time After Provisional Restorations. Int J Periodontics Restorative Dent 2019;39: 809-15. [8] Salama H, Salama M. The role of orthodontic extrusive remodeling in the enhancement of soft and hard tissue profiles prior to implant placement: a systematic approach to the management of extraction site defects. Int J Periodontics Restorative Dent1993;13,312-33. [9] Man Y, Wang Y, Qu Y, Wang P, Gong P. A palatal roll envelope technique for peri-implant mucosa reconstruction: a prospective case series study. Int J Oral Maxillofac Surg 2013;42:660-5. [10] Agarwal C, Deora S, Abraham D, Gaba R, Kumar BT,Kudva P. Vascularized interpositional periosteal connective tissue flap: A modern approach to augment soft tissue. J Indian Soc Periodontol 2015;19:72-7. [11] Man Y , Wu Q , Wang T , Gong P, Gong T , Qu Y. Split pedicle roll envelope technique around implants and pontics: a prospective case series study. Int J Oral Maxillofac Surg 2015;44:1295-301. [12] Urdaneta RA, Daher S, Lery J, Emanuel K, Chuang SK. Factors associated with crestal bone gain on single-tooth locking-taper implants: the effect of nonsteroidal anti-inflammatory drugs. Int J Oral Maxillofac Implants 2011;26, 1063-78. [13] De Rouck T, Eghbali R, Collys K, De Bruyn H, Cosyn J. The gingival biotype revisited: transparency of the periodontal probe through the gingival margin as a method to discriminate thin from thick gingiva. J Clin Periodontol 2009;36:,428-33. [14] Ronay V, Sahrmann P, Bindl A, Attin T, Schmidlin PR. Current status and perspectives of mucogingival soft tissue measurement methods. J Esthet Restor Dent 2011;23:146-56. [15] Mombelli A, Van Oosten MA, Schurch EJ, Lan NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol 1987;2:145-51. [16] Chang M, Wennström JL, Odman P, Andersson B. Implant supported single-tooth replacements compared to contralateral natural teeth. Crown and soft tissue dimensions. Clin Oral Implants Res 1999;10: 185-94. [17] Welander M, Abrahamsson I, Berglundh T. The mucosal barrier at implant abutments of different materials. Clin Oral Implants Res 2008;19:635-41. [18] Kajiwara N , Masaki C, Mukaibo T,Kondo Y, Nakamoto T, Hosokawa R. Soft tissue biological response to zirconia and metal implant abutments compared with natural tooth: microcirculation monitoring as a novel bioindicator. Implant Dent 2015;24:37-41. [19] Cooper LF, Ellner S, Moriarty J, Felton DA, Paquette D, Molina A, et al. Three-year evaluation of single-tooth implants restored 3 weeks after 1-stage surgery. Int J Oral Maxillofac Implants 2007;22:791-800. [20] Kan JY, Rungcharassaeng K, Liddelow G, Henry P, Goodacre CJ. Periimplant tissue response following immediate provisional restoration of scalloped implants in the esthetic zone: a one-year pilot prospective multicenter study. J Prosthet Dent 2007;97:109-18. [21] Al-Juboori MJ. Interdental Implant Papillae Grow up with Temporary Abutment displaced at Monthly Intervals. J Contemp Dent Pract 2015;16:422-6. [22] Finelle G, Papadimitriou D, Souza A, Katebi N,Gallucci G, Araújo M. Peri-implant soft tissue and marginal bone adaptation on implant with non-matching healing abutments: micro-CT analysis. Clin Oral Implants Res 2015;26:42-6. [23] Farronato D, Santoro G, Canullo L, Botticelli D, Maiorana C, Lang N. Establishment of the epithelial attachment and connective tissue adaptation to implants installed under the concept of
- [Derived] Luo W, Wang X, Chen Y, Hong Y, Qu Y, Man Y, Wu Y. Radiographic evaluation of a cross-shaped incision technique for thick-gingiva and thin-gingiva patients treated with implant-supported fixed prosthesis. BMC Oral Health. 2021 Dec 18;21(1):655. doi: 10.1186/s12903-021-02019-8. PMID 34922521